CLINICAL TRIAL: NCT06053151
Title: Cloud Platform Integration Model for Pregnant Women Exercise Consultation: Development, Construction and Evaluation
Brief Title: Cloud Platform Integration Model for Pregnant Women Exercise Consultation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, head of administion, Mackay Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MOST 111-2410-H-715 -001 -MY3
Record Dates: First submitted 2023-09-09; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Exercise; Pregnancy Related
Keywords: exercise counselling; pregnancy; women; platform; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiemental group (Experimental): The experimental group will receive the cloud platform integration model for exercise consultation intervention for two phases continue 24 weeks to promote exercise behavior during pregnancy.
  Interventions: Behavioral: exercise counselling
- control group (No Intervention): The control group will receive standard antenatal treatments without intervention.

INTERVENTIONS:
Behavioral: exercise counselling — . The experimental group will receive the cloud platform integration model for exercise consultation intervention for two phases continue 24 weeks to promote exercise behavior during pregnancy. The goal of the first phase was to start regular exercise, and the goal of the second phase was to continue regular exercise.
  Arms: experiemental group

SUMMARY:
To construct the platform for exercise counseling for pregnant women, and evaluate the effects of that telecare platform integration model for exercise consultation on exercise behaviors and prenatal health outcomes among pregnant women during pregnancy.

DETAILED DESCRIPTION:
This study will develop and construct an exercise counseling model with using cloud platform for women during pregnancy. In addition, we will evaluate the effects of that telecare platform integration model for exercise consultation on exercise behaviors and prenatal health outcomes among pregnant women during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women who less than 17 gestation and able to understand basic technologies such as smartphone and computer

Exclusion Criteria:

* women who had a diagnosis of pregnancy related compliactions and absolute limited exercise, such as preterm contraction, ruputer of menbrance, evidence of intrauterus growth retardation, heart and lung disease, cervical incompetence and/or medical conditions that influence exercise.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
increase physiacl activity | The data were collected before the intervention to childbirth: <16 week gestation, second trimester (24-26 weeks) and third trimester (34-36 weeks)
  measure by pregnancy physical activity questionnaire
decrese symptom distress | The data were collectedbefore the intervention to childbirth: <16 week gestation, second trimester (24-26 weeks) and third trimester (34-36 weeks)
  pregnancy related symptom distress scale
decrease pregnancy related complications | The data were collectedbefore the intervention to childbirth: <16 week gestation, second trimester (24-26 weeks) and third trimester (34-36 weeks)
  such as gestational diabetes, pregancy related hypertension, preclampsia, preterm labor.

SECONDARY OUTCOMES:
construct exercise counseling model | The data will be collected from pregnant women and experts perspectives; From date of first participant attend the focus group until the date of the last experts meeting , assessed up to 12 months
  intergrate the could platform in exercise counseling for pregnant women

CONTACTS AND LOCATIONS:
Overall Officials: Ching Fang Lee, PhD, Principal Investigator — Mackay Medical College

IPD SHARING:
Plan to Share IPD: No